CLINICAL TRIAL: NCT00468481
Title: Multi-Center, Randomized, Double-Blind Active-Controlled, Parallel Group Study to Investigate Plasma Folate, Red Blood Cell Folate and Homocysteine Levels During a 24 Week Oral Administration of an OC Containing Folate Compared to OC Alone
Brief Title: Efficacy and Safety Study for an Oral Contraceptive Containing Folate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91523; 310662 (Other: Company internal)
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Neural Tube Defects; Contraception; Oral Contraceptives (OC)
Keywords: Healthy women requesting contraception; Folic Acid
MeSH Terms: conditions — Neural Tube Defects | interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) (Experimental): 1 tablet 0.020 mg EE/3.0 mg DRSP/0.451 mg L-5-MTHF as calcium salt given orally/daily for 24 days followed by 1 tablet 0.451 mg L-5-MTHF as calcium salt given orally/daily for 4 days over a time period of 24 weeks
  Interventions: Drug: Drospirenone/Ethinylestradiol/Methyltetrahydrofolate
- Drospirenone (DRSP)/Ethinylestradiol (EE) (Active Comparator): 1 tablet 0.020 mg EE/3.0 mg DRSP [YAZ] given orally/daily for 24 days followed by 1 placebo tablet given orally/daily for 4 days over a time period of 24 weeks
  Interventions: Drug: Drospirenone/Ethinylestradiol (Yaz)

INTERVENTIONS:
Drug: Drospirenone/Ethinylestradiol/Methyltetrahydrofolate — 0.020 mg ethinylestradiol with 3.0 mg drospirenone and 0.451 mg L-5-methyltetrahydrofolate (L-5-MTHF)
  Arms: Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF)
Drug: Drospirenone/Ethinylestradiol (Yaz) — 0.020 mg ethinylestradiol with 3.0 mg drospirenone
  Arms: Drospirenone (DRSP)/Ethinylestradiol (EE)

SUMMARY:
The purpose of this study is to determine whether the study drug is safe and effective

DETAILED DESCRIPTION:
Acronym is used in result section: suspected/diagnosed (susp/diag)

ELIGIBILITY:
Inclusion Criteria:

- Healthy women between 18 and 40 requesting oral contraception

Exclusion Criteria:

- The use of steroidal oral contraceptives, or any drug that could alter Oral Contraception metabolism will be prohibited during the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 385 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (9):
  - Orange County Clinical Trials, Anaheim, California
  - Medical Center for Clinical Research, San Diego, California
  - SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - AAIPharma, Inc., Morrisville, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - NorthWest Kinetics, Tacoma, Washington

REFERENCES:
- [Result] Bart S Sr, Marr J, Diefenbach K, Trummer D, Sampson-Landers C. Folate status and homocysteine levels during a 24-week oral administration of a folate-containing oral contraceptive: a randomized, double-blind, active-controlled, parallel-group, US-based multicenter study. Contraception. 2012 Jan;85(1):42-50. doi: 10.1016/j.contraception.2011.05.013. Epub 2011 Jul 13. PMID 22067790
- [Result] Castano PM, Aydemir A, Sampson-Landers C, Lynen R. The folate status of reproductive-aged women in a randomised trial of a folate-fortified oral contraceptive: dietary and blood assessments. Public Health Nutr. 2014 Jun;17(6):1375-83. doi: 10.1017/S1368980013000864. Epub 2013 Mar 27. PMID 23534865
- [Result] Taylor TN, Farkouh RA, Graham JB, Colligs A, Lindemann M, Lynen R, Candrilli SD. Potential reduction in neural tube defects associated with use of Metafolin-fortified oral contraceptives in the United States. Am J Obstet Gynecol. 2011 Nov;205(5):460.e1-8. doi: 10.1016/j.ajog.2011.06.048. Epub 2011 Jun 21. PMID 21903192
- [Result] Campone M, Berton-Rigaud D, Joly-Lobbedez F, Baurain JF, Rolland F, Stenzl A, Fabbro M, van Dijk M, Pinkert J, Schmelter T, de Bont N, Pautier P. A double-blind, randomized phase II study to evaluate the safety and efficacy of acetyl-L-carnitine in the prevention of sagopilone-induced peripheral neuropathy. Oncologist. 2013;18(11):1190-1. doi: 10.1634/theoncologist.2013-0061. Epub 2013 Oct 8. PMID 24105751

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 572 subjects screened; 187 subjects screen failed; 385 subjects randomized
Period: Overall Study
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Started | 291 (6 of these randomized subjects did not take any study medication) | 94
Subjects Treated | 285 | 94
Completed | 203 | 70
Not Completed | 88 | 24
Not completed — Adverse Event | 13 | 3
Not completed — Lost to Follow-up | 25 | 8
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 18 | 8
Not completed — Withdrawal by Subject | 12 | 3
Not completed — susp/diag malignant/premalignant disease | 1 | 0
Not completed — Prohibited Medication | 1 | 1
Not completed — Egg Donor | 1 | 0
Not completed — Moved out of area | 4 | 1
Not completed — Non-Compliance | 5 | 0
Not completed — Other | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE) | Total
Number analyzed (Participants) | 285 | 94 | 379
Age, Continuous [Mean (Full Range); unit: years] | 24.8 [18 to 40] | 24.6 [18 to 39] | 24.7 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 94 | 379
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell (RBC) Folate Level at 24 Weeks
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: Week 24
Population: Analysis was based on Per Protocol Set (PPS) defined as all subjects who had no major protocol deviations and completed 24 weeks of treatment with valid data for one of the co-primary efficacy variables at baseline and week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 124 | 45
nmol/L | 1406.91 [1354.13 to 1459.68] | 1022.21 [934.6 to 1109.82]
Statistical Analysis 1: Comparison: Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) vs Drospirenone (DRSP)/Ethinylestradiol (EE); The null hypothesis was that the difference between DRSP/EE/MTHF and Yaz treatment groups in the RBC folate levels at week 24 was 0; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) with treatment as factor and Baseline (RBC folate) as covariate; Mean Difference (Final Values) = 384.70, 95% CI [282.42 to 486.98] — Difference = DRSP/EE/MTHF - YAZ

2. Primary Outcome: Plasma Folate Level at 24 Weeks
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 196 | 66
nmol/L | 60.55 [58.13 to 62.97] | 41.67 [37.50 to 45.85]
Statistical Analysis 1: Comparison: Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) vs Drospirenone (DRSP)/Ethinylestradiol (EE); The null hypothesis was that the difference between DRSP/EE/MTHF and Yaz treatment groups in the plasma folate levels at week 24 was 0; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) with treatment as factor and Baseline (plasma folate) as covariate; Mean Difference (Final Values) = 18.87, 95% CI [14.04 to 23.70] — Difference =DRSP/EE/MTHF - YAZ

3. Secondary Outcome: Mean Neural Tube Defect (NTD) Risk Reduction at Week 24
Description: The mean NTD risk reduction evaluated as the change from Baseline to Week 24 in NTD risk based on the formula of Daly et al (J Amer Med Assoc 1995;274(21):1698-702); NTD risk=exp (1.6463-1.2193 x natural log [RBC folate]) where natural log [RBC folate] is the natural log of RBC folate measured in nmol/L; Change from Baseline to Week 24 in NTD risk=NTD risk at Week 24 - NTD risk at Baseline
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per 1000 birth
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 124 | 45
per 1000 birth | -0.51 (0.41) | -0.03 (0.26)

4. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Folate Levels at Week 4
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: baseline and up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 125 | 43
nmol/L | 110.9 (207.28) | -37.6 (195.88)

5. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Folate Levels at Week 8
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: baseline and up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 122 | 43
nmol/L | 310.3 (231.47) | 68.2 (155.26)

6. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Folate Levels at Week 12
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: baseline and up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 127 | 41
nmol/L | 405.8 (243.88) | 86.5 (177.81)

7. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Folate Levels at Week 16
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: baseline and up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 120 | 46
nmol/L | 448.9 (280.37) | 68.0 (186.44)

8. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Folate Levels at Week 20
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: baseline and up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 123 | 44
nmol/L | 452.7 (284.64) | 64.6 (194.89)

9. Secondary Outcome: Mean Change From Baseline in Plasma Folate Levels at Week 4
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: baseline and up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 192 | 65
nmol/L | 15.2 (22.07) | 0.6 (14.29)

10. Secondary Outcome: Mean Change From Baseline in Plasma Folate Levels at Week 8
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: baseline and up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 193 | 66
µg/L | 18.4 (19.17) | 2.2 (14.63)

11. Secondary Outcome: Mean Change From Baseline in Plasma Folate Levels at Week 12
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: baseline and up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 194 | 66
nmol/L | 17.6 (20.1) | 0.3 (15.24)

12. Secondary Outcome: Mean Change From Baseline in Plasma Folate Levels at Week 16
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: baseline and up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 194 | 65
nmol/L | 17.6 (12.43) | 2.4 (16.44)

13. Secondary Outcome: Mean Change From Baseline in Plasma Folate Levels at Week 20
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: baseline and up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 193 | 66
nmol/L | 15.1 (22.71) | -1.6 (15.65)

14. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 4
Description: Homocysteine concentrations in plasma were determined by Fluorescence Polarization Immunoassays (FPIA) using the Abbot AxSym analyzer in a clinical laboratory setting.
Time Frame: baseline and up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 194 | 65
µg/L | 0 (1.04) | 0 (0.69)

15. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 8
Description: as for outcome 14
Time Frame: baseline and up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 195 | 66
µg/L | -0.2 (0.9) | 0 (1)

16. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 12
Description: as for outcome 14
Time Frame: baseline and up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 196 | 66
µg/L | -0.3 (1.07) | 0 (0.93)

17. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 16
Description: as for outcome 14
Time Frame: baseline and up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 194 | 65
µg/L | -0.2 (1.02) | -0.1 (0.93)

18. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 20
Description: as for outcome 14
Time Frame: baseline and up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 195 | 66
µg/L | -0.2 (1.07) | -0.2 (0.91)

19. Secondary Outcome: Mean Change From Baseline in Plasma Homocysteine Levels at Week 24
Description: as for outcome 14
Time Frame: baseline and up to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 195 | 66
µg/L | -0.3 (0.93) | 0.1 (1.24)

20. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Baseline
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: at baseline (week 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 90 | 40
nmol/L | 910.9 (276.05) | 915.1 (233.97)

21. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Baseline
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: at baseline (week 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 54 | 12
nmol/L | 1122.8 (504.7) | 1345.0 (301.76)

22. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 4
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 80 | 35
nmol/L | 1007.1 (329.67) | 889.5 (262.42)

23. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 4
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 50 | 9
nmol/L | 1175.7 (428.58) | 1256.1 (190.89)

24. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 8
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 76 | 33
nmol/L | 1184.8 (338.5) | 970.4 (252.79)

25. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 8
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 50 | 10
nmol/L | 1412.7 (436.69) | 1407.6 (290.18)

26. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 12
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 79 | 33
nmol/L | 1308.9 (374.61) | 1025.2 (287.55)

27. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 12
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 50 | 10
nmol/L | 1469.8 (454.62) | 1378.4 (375.15)

28. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 16
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 76 | 35
nmol/L | 1365.2 (403.12) | 967.6 (255.78)

29. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 16
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 50 | 11
nmol/L | 1460.5 (472.23) | 1454.7 (355.5)

30. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 20
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 78 | 33
nmol/L | 1419.8 (558.1) | 981.3 (252.85)

31. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 20
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 49 | 13
nmol/L | 1486.6 (462.8) | 1435.9 (319.33)

32. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 24
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 87 | 37
nmol/L | 1355.3 (364.85) | 949.2 (256.26)

33. Post Hoc Outcome: Mean Red Blood Cell (RBC) Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 24
Description: RBC folate=([whole blood folate*100]-[plasma folate*(100-hematocrit)])/hematocrit
Time Frame: up to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 51 | 10
nmol/L | 1500.3 (525.71) | 1316.1 (237.44)

34. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Baseline
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: at baseline (week 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 120 | 47
nmol/L | 41.7 (16.2) | 41.5 (15.57)

35. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Baseline
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: at baseline (week 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 76 | 19
nmol/L | 50.3 (18.45) | 47.1 (17.3)

36. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 4
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 119 | 47
nmol/L | 59.6 (24.83) | 43.1 (17.98)

37. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 4
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 73 | 18
nmol/L | 60.4 (27.56) | 45.9 (21.19)

38. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 8
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 118 | 47
nmol/L | 60.8 (22.41) | 41.8 (14.96)

39. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 8
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 75 | 19
nmol/L | 68.1 (26.60) | 54.1 (30.16)

40. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 12
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 119 | 47
nmol/L | 59.5 (20.39) | 42.3 (17.19)

41. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 12
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 75 | 19
nmol/L | 67.4 (23.69) | 46.4 (17.55)

42. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 16
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 118 | 46
nmol/L | 59.4 (18.89) | 43.2 (18.4)

43. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 16
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 76 | 19
nmol/L | 67.5 (26.38) | 51.8 (21.08)

44. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 20
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 118 | 47
nmol/L | 59.8 (21.11) | 39.7 (16.74)

45. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 20
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 75 | 19
nmol/L | 61.5 (24.16) | 45.9 (14.54)

46. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (Without Additional Folate Supplementation) at Week 24
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 120 | 47
nmol/L | 58.7 (17.73) | 39.8 (18.02)

47. Post Hoc Outcome: Mean Plasma Folate Levels by Additional Folate Supplementation (With Additional Folate Supplementation) at Week 24
Description: Folate concentrations in plasma were determined by an appropriately validated microbiological assay.
Time Frame: up to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Number analyzed (Participants) | 76 | 19
nmol/L | 64.0 (22.61) | 43.7 (16.5)

ADVERSE EVENTS:
Arm/Group | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) | Drospirenone (DRSP)/Ethinylestradiol (EE)
Serious Adverse Events (participants affected / at risk) | 3/285 | 0/94
Other Adverse Events (participants affected / at risk) | 103/285 | 44/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) (N=285) | Drospirenone (DRSP)/Ethinylestradiol (EE) (N=94)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Human papilloma virus test positive (Investigations) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drospirenone (DRSP)/Ethinylestradiol (EE)/Metafolin (MTHF) (N=285) | Drospirenone (DRSP)/Ethinylestradiol (EE) (N=94)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 6 (6) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (11) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 9 (9) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 30 (32) | 9 (10)
Urinary tract infection (Infections and infestations) | 10 (11) | 2 (2)
Blood cholinesterase decreased (Investigations) | 1 (1) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2)
Low density lipoprotein increased (Investigations) | 17 (17) | 8 (8)
Prothrombin level decreased (Investigations) | 0 (0) | 2 (2)
Human papilloma virus test positive (Investigations) | 10 (10) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 6 (9) | 4 (6)
Migraine (Nervous system disorders) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Cervical dysplasia (Reproductive system and breast disorders) | 10 (10) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less